CLINICAL TRIAL: NCT01787591
Title: Dairy Fat as a Mediator of Vitamin E Adequacy in Individuals With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Associate Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012H0344
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-09

CONDITIONS: Non-alcoholic Fatty Liver; Metabolic Syndrome
Keywords: Vitamin E; Metabolic syndrome; Liver disease; Non-alcoholic liver steatohepatitis; Fatty liver; Dairy consumption
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Liver Diseases; Fatty Liver | interventions — Diet, Fat-Restricted; Soy Milk

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acute Fat-Free Milk Ingestion (Experimental): Participants will ingest 1 cup of fat-free milk with 15 mg deuterium-labeled alpha-tocopherol.
  Interventions: Other: Fat-Free Milk
- Acute Low-Fat Milk Ingestion (Experimental): Participants will ingest 1 cup of low-fat milk with 15 mg deuterium-labeled alpha-tocopherol.
  Interventions: Other: Low-Fat Milk
- Acute Full-Fat Milk Ingestion (Experimental): Participants will ingest 1 cup of full-fat milk with 15 mg deuterium-labeled alpha-tocopherol.
  Interventions: Other: Full-Fat Milk
- Acute Soy Milk Ingestion (Experimental): Participants will ingest 1 cup of soy milk with 15 mg deuterium-labeled alpha-tocopherol.
  Interventions: Other: Soy Milk

INTERVENTIONS:
Other: Fat-Free Milk — Fat-free milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
  Arms: Acute Fat-Free Milk Ingestion
Other: Low-Fat Milk — Low-fat milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
  Arms: Acute Low-Fat Milk Ingestion
Other: Full-Fat Milk — Full-fat milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
  Arms: Acute Full-Fat Milk Ingestion
Other: Soy Milk — Soy milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
  Arms: Acute Soy Milk Ingestion

SUMMARY:
This study is conducted to investigate if vitamin E status in healthy individuals and individuals with metabolic syndrome can be improved by dairy fat. The investigators hypothesize that full-fat dairy will substantially increase the bioavailability of alpha-tocopherol, a form of vitamin E. The results of this study will contribute to the application of dairy fat as a simple and effective strategy for improving vitamin E status, which is partly due to poor vitamin E intake. By completing this study, the investigators anticipate developing new dietary recommendations to achieve adequate vitamin E status through the regular consumption of dairy fat paired with foods containing vitamin E.

DETAILED DESCRIPTION:
Nonalcoholic steatohepatitis (NASH) is the hepatic manifestation of metabolic syndrome and affects >70 million Americans. Weight loss and vitamin E supplementation are leading strategies for preventing and/or treating NASH. However, the long-term success of weight loss is limited and >92% of Americans fail to meet dietary recommendations for vitamin E. Thus, the objective is to define the extent to which dairy fat facilitates adequate vitamin E status in individuals with metabolic syndrome, a population at high-risk for NASH, by improving α-tocopherol bioavailability. The central hypothesis is that full-fat dairy will substantially increase alpha-tocopherol (a-T) bioavailability to the extent needed to facilitate production of alpha-carboxyethyl-hydroxy-chromanol (a-CEHC), a metabolite of a-T that predict a-T status. The will therefore complete the following specific aims: 1) define milk fat-mediated improvements in a-T bioavailability, and 2) define dairy fat-mediated improvements in a-T status. This study involves a randomized crossover study design where healthy adults and those with metabolic syndrome (n = 10/group) will ingest deuterium-labeled a-T (15 mg) with 1 cup of either fat-free milk, low-fat milk, whole milk, or soy milk. Urine and blood samples will be collected at timed intervals prior to and following milk consumption. Blood will be collected at timed intervals over 72 h, and plasma will be analyzed by liquid chromatography with mass spectrometry to determine pharmacokinetic parameters by measuring labeled and unlabeled a-T and a-CEHC. Risk to participants is expected to be minimal and will be outlined in the informed consent form in clear and simple terms. Upon successful completion of this study, it is expected to show that a-T bioavailability increases in a milk fat-dependent manner and that dairy milk compared with soy milk significantly improves a-T bioavailability. The results are expected to provide timely evidence demonstrating the amount and type of fat needed to achieve optimal vitamin E status specifically in a population of significant public health concern. Overall, these studies will fill a substantial knowledge gap regarding the importance of dairy fat in contributing to optimal health and provide a simple dietary approach to ameliorate poor vitamin E status among a significant proportion of Americans.

ELIGIBILITY:
Inclusion Criteria:

* specific criteria of the metabolic syndrome: large waist circumference (>102 or >89 cm for men and women, respectively), high fasting triglycerides (150-300 mg/dL), low fasting HDL (<40 and <50 mg/dL for men and women, respectively), high blood pressure (>130/85 mm Hg) and high fasting glucose (110-180 mg/dL)
* BMI: >30 kg/m2,
* non-dietary supplement users for >2-mo
* no use of medications known to affect lipid metabolism
* no history of gastrointestinal disorders
* resting blood pressure <140 mm Hg
* not taking any medications that control hypertension

Exclusion Criteria:

* lactose-intolerance
* excessive alcohol consumption (>3 drinks/d)
* >5 h/wk of aerobic activity
* women who are pregnant, lactating, or have initiated or changed birth control in the past 3-mo
* plasma alpha-tocopherol >20 μmol/L.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared when it becomes available

REFERENCES:
- [Result] Mah E, Sapper TN, Chitchumroonchokchai C, Failla ML, Schill KE, Clinton SK, Bobe G, Traber MG, Bruno RS. alpha-Tocopherol bioavailability is lower in adults with metabolic syndrome regardless of dairy fat co-ingestion: a randomized, double-blind, crossover trial. Am J Clin Nutr. 2015 Nov;102(5):1070-80. doi: 10.3945/ajcn.115.118570. Epub 2015 Oct 7. PMID 26447154
- [Derived] Traber MG, Mah E, Leonard SW, Bobe G, Bruno RS. Metabolic syndrome increases dietary alpha-tocopherol requirements as assessed using urinary and plasma vitamin E catabolites: a double-blind, crossover clinical trial. Am J Clin Nutr. 2017 Mar;105(3):571-579. doi: 10.3945/ajcn.116.138495. Epub 2017 Jan 11. PMID 28077381

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Fat-Free Milk Ingestion First: Participants ingested fat-free milk first and then the remaining three milks in a randomized order: low-fat milk, full-fat milk, and soy milk.
  Participants will ingest 1 cup of fat-free milk with 15 mg deuterium-labeled alpha-tocopherol.
  Fat-Free Milk: Fat-free milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
- Acute Low-Fat Milk Ingestion First: Participants ingested low-free milk first and then the remaining three milks in a randomized order: fat-fat milk, full-fat milk, and soy milk.
  Participants will ingest 1 cup of low-fat milk with 15 mg deuterium-labeled alpha-tocopherol.
  Low-Fat Milk: Low-fat milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
- Acute Full-Fat Milk Ingestion First: Participants ingested full-free milk first and then the remaining three milks in a randomized order: low-fat milk, low-fat milk, and soy milk.
  Participants will ingest 1 cup of full-fat milk with 15 mg deuterium-labeled alpha-tocopherol.
  Full-Fat Milk: Full-fat milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
- Acute Soy Milk Ingestion First: Participants ingested soy milk first and then the remaining three milks in a randomized order: low-fat milk, full-fat milk, and fat-free milk.
  Participants will ingest 1 cup of soy milk with 15 mg deuterium-labeled alpha-tocopherol.
  Soy Milk: Soy milk ingestion with 15 mg deuterium-labeled alpha-tocopherol.
Period: Period 1 (Cross-over Arm 1)
Arm/Group | Acute Fat-Free Milk Ingestion First | Acute Low-Fat Milk Ingestion First | Acute Full-Fat Milk Ingestion First | Acute Soy Milk Ingestion First
Started | 5 | 5 | 5 | 6
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Period 2 (Cross-over Arm 2)
Arm/Group | Acute Fat-Free Milk Ingestion First | Acute Low-Fat Milk Ingestion First | Acute Full-Fat Milk Ingestion First | Acute Soy Milk Ingestion First
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 (Cross-over Arm 3)
Arm/Group | Acute Fat-Free Milk Ingestion First | Acute Low-Fat Milk Ingestion First | Acute Full-Fat Milk Ingestion First | Acute Soy Milk Ingestion First
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 4 (Cross-over Arm 4)
Arm/Group | Acute Fat-Free Milk Ingestion First | Acute Low-Fat Milk Ingestion First | Acute Full-Fat Milk Ingestion First | Acute Soy Milk Ingestion First
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Participants; Metabolic Syndrome Participants: As a randomized crossover study design, participants were stratified by health status (healthy versus metabolic syndrome) and received fat-free milk, low-fat milk, full-fat milk, and soy milk in a randomized order.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Metabolic Syndrome Participants | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (4) | 32.8 (5.1) | 31.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 22.6 (2.2) | 37.7 (9.4) | 30.2 (10.2)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 89.2 (6.2) | 107.6 (4.2) | 98.4 (13.9)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118.8 (9.5) | 128.2 (23.6) | 123.5 (18.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.0 (7.9) | 79.0 (10.1) | 76.5 (9.2)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 75.2 (6.5) | 116.1 (23.7) | 95.7 (27.0)
Triglyceride [Mean (Standard Deviation); unit: mg/dL] | 82.0 (30.4) | 152.7 (68.1) | 117.4 (62.8)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 56.0 (9.9) | 41.2 (10.8) | 48.6 (12.6)
alpha-tocopherol [Mean (Standard Deviation); unit: umol/L] | 22.2 (3.9) | 23.9 (2.8) | 23.1 (3.4)
alpha-tocopherol [Mean (Standard Deviation); unit: umol/mmol lipid] | 4.54 (0.85) | 3.71 (0.85) | 4.13 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0-72 h (Deuterium Labeled Alpha-tocopherol)
Time Frame: 0, 3, 6, 9, 12, 24, 36, 48, and 72 h post test meal
Measure: Mean (Standard Error); unit: umol/L x h
Groups:
- Acute Soy Milk Ingestion: Participants received 1 cup of soy milk with deuterium labeled alpha-tocopherol
Arm/Group | Acute Fat-Free Milk Ingestion | Acute Low-Fat Milk Ingestion | Acute Full-Fat Milk Ingestion | Acute Soy Milk Ingestion
Number analyzed (Participants) | 20 | 20 | 20 | 20
umol/L x h
  Healthy Participants | 103 (7) | 115 (8) | 102 (8) | 102 (5)
  Metabolic Syndrome Participants | 86 (8) | 84 (7) | 81 (7) | 74 (11)

2. Primary Outcome: Cmax
Description: Maximal plasma concentration of deuterium labelled alpha-tocopherol
Time Frame: 0-72 h post-meal
Measure: Mean (Standard Error); unit: umol/L
Groups:
- Acute Soy Milk Ingestion: Participants ingested 1 cup of soy milk with deuterium labeled alpha-tocopherol
Arm/Group | Acute Fat-Free Milk Ingestion | Acute Low-Fat Milk Ingestion | Acute Full-Fat Milk Ingestion | Acute Soy Milk Ingestion
Number analyzed (Participants) | 20 | 20 | 20 | 20
umol/L
  Healthy | 2.67 (0.2) | 2.98 (0.18) | 2.55 (0.21) | 2.67 (0.13)
  Metabolic Syndrome | 2.14 (0.2) | 2.01 (0.19) | 1.98 (0.16) | 1.88 (0.27)

3. Primary Outcome: Tmax
Description: Time to maximal plasma concentration of deuterium labelled alpha-tocopherol
Time Frame: 0-72 h post-meal
Measure: Mean (Standard Error); unit: h
Arm/Group | Acute Fat-Free Milk Ingestion | Acute Low-Fat Milk Ingestion | Acute Full-Fat Milk Ingestion | Acute Soy Milk Ingestion
Number analyzed (Participants) | 20 | 20 | 20 | 20
h
  Healthy | 12 (0) | 12 (0) | 13.2 (1.2) | 12 (0)
  Metabolic Syndrome | 12 (0) | 12 (0) | 12 (0) | 12 (0)

4. Primary Outcome: Elimination Rate
Description: Rate of plasma elimination of deuterium labelled alpha-tocopherol
Time Frame: 0-72 h post-meal
Measure: Mean (Standard Error); unit: mmol/L/h
Arm/Group | Acute Fat-Free Milk Ingestion | Acute Low-Fat Milk Ingestion | Acute Full-Fat Milk Ingestion | Acute Soy Milk Ingestion
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmol/L/h
  Healthy | 0.022 (0.001) | 0.024 (0.001) | 0.023 (0.001) | 0.023 (0.001)
  Metabolic Syndrome | 0.019 (0.001) | 0.020 (0.001) | 0.021 (0.001) | 0.022 (0.001)

5. Primary Outcome: Estimated Absorption (% Dose)
Description: Absorption of deuterium labelled alpha-tocopherol
Time Frame: 0-72 h post-meal
Measure: Mean (Standard Error); unit: % dose
Arm/Group | Acute Fat-Free Milk Ingestion | Acute Low-Fat Milk Ingestion | Acute Full-Fat Milk Ingestion | Acute Soy Milk Ingestion
Number analyzed (Participants) | 20 | 20 | 20 | 20
% dose
  Healthy | 27.8 (1.4) | 32.4 (1.6) | 28.4 (1.3) | 28.1 (0.88)
  Metabolic Syndrome | 26.6 (1.8) | 26.0 (2.5) | 25.6 (1.9) | 24.62 (2.72)

ADVERSE EVENTS:
Arm/Group | Acute Fat-Free Milk Ingestion | Acute Low-Fat Milk Ingestion | Acute Full-Fat Milk Ingestion | Acute Soy Milk Ingestion
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No